CLINICAL TRIAL: NCT04282460
Title: A Randomized Clinical Trial of Ba Duan Jin in Treatment of Attention Deficit Hyperactivity Disorder With Hyperactive-Impulsive Symptom
Brief Title: Ba Duan Jin in Treatment of Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19401931200
Record Dates: First submitted 2020-02-21; First posted 2020-02-24 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Chinese traditional medicine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The present study will be carried out using a parallel randomized study design. Each participant will be randomly assigned either to the Baduanjin intervention or to the regular physical exercise control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The medical treatment of participants will be given by a doctor who does not know the study group of the patient. The investigator of the primary outcome and secondary outcome will also be unaware of the grouping of the patient. One psychiatrist blind of grouping will ask parents about the ADHD Hyperactivity/Impulsivity symptom of their children and rate it with SNAP-IV Hyperactivity/Impulsivity score. Another Chinese traditional medical doctor blind of grouping will evaluate the severity of traditional Chinese medicine symptoms of children and rate it with TCM symptom scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin practice (Experimental): Baduanjin practice group will be asked to use the Baduanjin training system to practice the whole set of Baduanjin at least once a day and at least 5 days each week for 3 months.
  Interventions: Behavioral: Baduanjin practice
- Regular physical exercise (Active Comparator): The regular physical exercise group will be asked to take physical exercise for at least half an hour every day in addition to regular physical activities at school.
  Interventions: Behavioral: Regular physical exercise

INTERVENTIONS:
Behavioral: Baduanjin practice — Use the Baduanjin training system to practice the whole set of Baduanjin at least once a day and at least 5 days each week for 3 months.
  Arms: Baduanjin practice
Behavioral: Regular physical exercise — Take physical exercise for at least half an hour every day in addition to regular physical activities at school.
  Arms: Regular physical exercise

SUMMARY:
This study is designed to test if Baduanjin training can reduce the hyperactive-impulsive symptoms of children with Attention deficit hyperactivity disorder (ADHD) compared to routine excise. Investigators will also evaluate if the Baduanjin training will positively affect Chinese Traditional Medicine (TCM) symptoms compared to controls and if these impacts are related to the change of the executive function.

DETAILED DESCRIPTION:
ADHD is a common neurodevelopmental disorder characterized by a persistent pattern of inattention and/or hyperactivity and impulsivity, resulting in functional impairment in multiple settings. The prevalence in China is estimated to be 6.26%. From the point of Chinese Traditional Medicine (TCM), ADHD can be divided into 4 categories according to the symptom differentiation in TCM.

Aerobic exercise is known to improve executive function (EF) performance, which is known as the core deficit of ADHD, therefore reduce ADHD symptoms. Aerobic exercise with the component of self-control and development of character is reported to improve EF.

Baduanjin is one of the aerobic exercises that has been handed down since the northern song dynasty, serving as Chinese physical and breathing exercises. The eight movements of Baduanjin are required to be gentle, slow, elastic and appropriate which not only require the practitioner to control physical activity but also require a combination of cognitive activities. Researchers found that Baduanjin has a positive protective effect on cognitive function such as selective attention in patients with mild cognitive impairment adults.

Therefore, investigators designed the Baduanjin training system. This is a combination of a physical and cognitive training program and a video game with a motivation system, interesting and engaging for children with ADHD to practice on.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ADHD, Combined Presentation or Predominantly Hyperactive-Impulsive Presentation
* Doctor rated SNAP-IV Hyperactivity/Impulsivity score≥12
* Full-Scale Intelligence Quotient>=80 (Wechsler intelligence scale for children-IV)
* Resident in Shanghai，Zhejiang province and Jiangsu province, parents and children agree to participate in the intervention

Exclusion Criteria:

* Using psychiatric medication other than methylphenidate
* Attending any other type of regular physical exercises except the gym class in school during the intervention period
* Accepting any type of psychological treatment during the intervention
* Comorbid with epileptic disorder or other existing physical disorder, Tourette syndrome, Autism Spectrum Disorder, learning disorder, mood disorder, psychiatric disorder, or under suicidal risk
* Attending any other clinical research at the same time

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2020-10-24 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Hyperactivity/Impulsivity score change in SNAP-IV scale | Baseline, 3 months after enrollment
  The Swanson, Nolan, and Pelham Questionnaire (SNAP-IV) Rating Scale is a revised version of the Swanson, Nolan and Pelham (SNAP) Questionnaire that utilizes the DSM-IV criteria for ADHD and oppositional defiant disorder, rated by caregiver or professionals. It comprises three subscales: Inattention, Hyperactivity/Impulsivity, and Oppositional Defiant Disorder. The score of each item is rated with a 4-point Likert scale (0 = not at all, 3 = very much). We choose the 9-item-Hyperactivity/Impulsivity subscale for the evaluation of change in ADHD Hyperactivity/Impulsivity symptom in children. The score of Hyperactivity/Impulsivity subscale is calculated by adding the 9 items, the score will range from 0 to 27. The change of score is calculated by Hyperactivity/Impulsivity score at 3 months enrollment (both Baduanjin practice group and Regular physical exercise group went through 3 months of intervention at this point) minus Hyperactivity/Impulsivity score at baseline (enrollment).

SECONDARY OUTCOMES:
Change of Scoring evaluation of the TCM symptoms | Baseline, 3 months after enrollment
  The TCM symptom scale was developed from the guideline system for traditional Chinese medicine new drug clinical research to evaluate the severity of TCM symptoms of children. This scale include 23 items, each presents one common TCM symptom. Each symptom is rated 1-4 points according to its severity. The total score is calculated by adding the scores of all 23 items. The change of score is calculated by TCM symptoms score after 3 months of enrollment (both Baduanjin practice group and Regular physical exercise group went through 3 months of intervention at this point) minus TCM symptoms score at baseline (enrollment).

CONTACTS AND LOCATIONS:
Overall Officials: Daqian Zhu, PhD, Study Chair — Department of Psychological Medicine, Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davis CL, Tomporowski PD, McDowell JE, Austin BP, Miller PH, Yanasak NE, Allison JD, Naglieri JA. Exercise improves executive function and achievement and alters brain activation in overweight children: a randomized, controlled trial. Health Psychol. 2011 Jan;30(1):91-8. doi: 10.1037/a0021766. PMID 21299297
- [Background] Drollette ES, Scudder MR, Raine LB, Moore RD, Saliba BJ, Pontifex MB, Hillman CH. Acute exercise facilitates brain function and cognition in children who need it most: an ERP study of individual differences in inhibitory control capacity. Dev Cogn Neurosci. 2014 Jan;7:53-64. doi: 10.1016/j.dcn.2013.11.001. Epub 2013 Nov 16. PMID 24309300
- [Background] Pontifex MB, Saliba BJ, Raine LB, Picchietti DL, Hillman CH. Exercise improves behavioral, neurocognitive, and scholastic performance in children with attention-deficit/hyperactivity disorder. J Pediatr. 2013 Mar;162(3):543-51. doi: 10.1016/j.jpeds.2012.08.036. Epub 2012 Oct 17. PMID 23084704
- [Background] Verburgh L, Konigs M, Scherder EJ, Oosterlaan J. Physical exercise and executive functions in preadolescent children, adolescents and young adults: a meta-analysis. Br J Sports Med. 2014 Jun;48(12):973-9. doi: 10.1136/bjsports-2012-091441. Epub 2013 Mar 6. PMID 23467962

DOCUMENTS (2):
  • Study Protocol (2022-11-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT04282460/Prot_001.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT04282460/SAP_000.pdf